CLINICAL TRIAL: NCT00682474
Title: School Nurse-Delivered Smoking Cessation Intervention
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Lori Pbert, Professor of Medicine, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01CA114556 (NIH)
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-08

CONDITIONS: Cigarette Smoking; Nicotine Dependence
Keywords: Cigarette smoking; Nicotine dependence; Adolescents; Youth; School health; Randomized controlled trial
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use Disorder | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CI (Experimental): Four 30-minute individual student-centered smoking cessation counseling intervention sessions delivered by school nurses to adolescent smokers in grades 9-12
  Interventions: Behavioral: Counseling Intervention
- II (Active Comparator): Attention-control comparison condition consisting of four individual sessions with the school nurse to check smoking status and deliver a series of standardized pamphlets on smoking and cessation to adolescent smokers in grades 9-12
  Interventions: Behavioral: Information Intervention

INTERVENTIONS:
Behavioral: Counseling Intervention — Four 30-minute individual student-centered smoking cessation counseling intervention sessions delivered by school nurses to adolescent smokers in grades 9-12
  Other Names: Calling It Quits
  Arms: CI
Behavioral: Information Intervention — Attention-control comparison condition consisting of four individual sessions with the school nurse to check smoking status and deliver a series of standardized pamphlets on smoking and cessation to adolescent smokers in grades 9-12
  Arms: II

SUMMARY:
The purpose of this study is to conduct a randomized controlled school-based trial to evaluate the effectiveness of a four-session school nurse-delivered smoking cessation intervention in increasing abstinence rates among high school students who smoke.

DETAILED DESCRIPTION:
Smoking is the largest preventable cause of disease and premature death in the United States. Adolescent smoking is the greatest predictor of adult smoking and is associated with adverse health effects during adolescence. Twenty-two percent of high school students report current smoking (past 30 days). As the primary health professional in the school setting, school nurses have a tremendous opportunity to play a key role in treating adolescent smokers. A randomized controlled trial (RCT) conducted by the investigators in 71 high schools in Massachusetts demonstrated the feasibility of school nurses delivering a four-session individual counseling intervention to adolescents who want to stop smoking and its potential efficacy in increasing self-reported short term (6-week and 3-month) quit rates. Although promising, the preliminary study lacked biochemical validation and long-term follow-up on the maintenance of the intervention effects, and was conducted with a primarily white student population. This application seeks to evaluate the effectiveness of the intervention using a more rigorous methodology, including biochemical validation of self-reported smoking behavior and longer-term follow-up (6 and 12 months post-intervention), a study design that compares the intervention to an information only attention-control condition, and recruitment from ethnically diverse schools to increase the generalizability of our findings.

The overall aim of the proposed study is to conduct a randomized controlled school-based trial (RCT) to evaluate the effectiveness of a school nurse-delivered smoking cessation intervention in increasing 30 day abstinence rates among high school students who smoke. Forty high schools serving a diverse student population will be recruited and randomly assigned to one of two conditions: (1) Special Intervention (SI) - four 30-minute individual patient-centered smoking cessation counseling intervention sessions based on the Public Health Service (PHS) clinical practice guideline delivered by school nurses; or (2) Information Only (IO) attention-control comparison condition - four individual sessions with the school nurse to check smoking status and deliver a standardized series of informational pamphlets on smoking and cessation. Participant assessments will occur at study entry (baseline) and at 3-,12-month follow-up. Thirty students enrolled in grades 9 through 12 who report smoking within the past 30 days and willingness to participate in a smoking cessation intervention study will be recruited from each school (n=1200) to provide 25 completed assessments per school at 12-month follow-up (n=1000). If found effective, the study products (i.e., intervention protocol, student materials, training manual, and estimated costs of intervention implementation) will facilitate dissemination of the intervention to school nurses nationally.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in grades 9-12
* report smoking at least one puff of a cigarette in the past 30 days
* willingness to participate in a smoking cessation intervention study
* able to speak and read English
* able to complete the baseline questionnaire independently, indicating ability to complete study assessments and protocols
* intending to remain enrolled in the school for the remainder of the school year
* willing to provide contact information for the next 12 months

Exclusion Criteria:

* unwilling/unable to provide informed assent
* planning to move out of the area in the next 6 months

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1058 (Actual)
Dates: Start 2006-09; Primary Completion 2009-06 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Abstinence from cigarette smoking in the past 30 days at 3 months and 1 year. | 3 months and 1 year post baseline

SECONDARY OUTCOMES:
Reduction in number of cigarettes and days smoked | 3 months and 1 year post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Lori Pbert, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] Pbert L, Druker S, DiFranza JR, Gorak D, Reed G, Magner R, Sheetz AH, Osganian S. Effectiveness of a school nurse-delivered smoking-cessation intervention for adolescents. Pediatrics. 2011 Nov;128(5):926-36. doi: 10.1542/peds.2011-0520. Epub 2011 Oct 17. PMID 22007015